CLINICAL TRIAL: NCT02805439
Title: Efficacy and Safety of S 47445 Versus Placebo as Adjunctive Treatment of Major Depressive Disorder in Patients With an Inadequate Response to Antidepressant Therapy: A Randomised, Double-blind, Placebo Controlled International, Multicentre Study
Brief Title: Efficacy and Safety of S 47445 Versus Placebo as Adjunctive Treatment in Depressed Patients Not Fully Recovered From Depressive Symptoms With a Current Antidepressant Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR Association (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL2-47445-014; 2015-003867-13 (EudraCT Number)
Record Dates: First submitted 2016-06-13; First posted 2016-06-20 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- S47445 15mg (Experimental)
  Interventions: Drug: S47445 15mg
- S47445 50mg (Experimental)
  Interventions: Drug: S47445 50mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S47445 15mg — One tablet of S47445 15 mg taken orally once a day during breakfast concomitantly to the current selective serotonin reuptake inhibitor treatment, starting the day after inclusion visit and ending the day of the W8 visit.
  Arms: S47445 15mg
Drug: S47445 50mg — One tablet of S47445 50 mg taken orally once a day during breakfast concomitantly to the current selective serotonin reuptake inhibitor treatment, starting the day after inclusion visit and ending the day of the W8 visit.
  Arms: S47445 50mg
Drug: Placebo — One tablet of placebo taken orally once a day during breakfast concomitantly to the current selective serotonin reuptake inhibitor treatment, starting the day after inclusion visit and ending the day of the W8 visit.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of S47445 versus placebo as adjunctive treatment of Major Depressive Disorder in patients with an inadequate response to antidepressant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Fulfilling DSM-5 criteria for Major Depressive Disorder confirmed by the brief structured interview M.I.N.I. (single or recurrent episode, current episode ≤ 12 months, current depressive episode of moderate or severe intensity, with or without anxious distress, with or without melancholic features, without mixed features or atypical features, without seasonal pattern, without psychotic features, without catatonic features, without peripartum onset for the current episode)
* Patients treated for the current depressive episode with an antidepressant treatment with SSRI (fluoxetine, citalopram, paroxetine, escitalopram or sertraline) given in monotherapy at recommended dose for at least 6 weeks and no more than 4 months and with a stable dosage for at least 3 weeks
* HAM-D total score ≥ 20
* Clinical Global Impression Severity of illness (item 1): 6 ≥ CGI-S ≥ 4
* Antidepressant Treatment Response Questionnaire (ATQR) < 50% for the current SSRI
* Absence of any abnormalities likely to interfere with the conduct of the study (ECG, vital signs, laboratory tests, medical history)

Exclusion Criteria:

* Depressive episode of mild intensity according to DSM-5 criteria
* All types of depressive episodes other than those occurring in a Major Depressive Disorder (Persistent Depressive Disorder (Dysthymia) according to DSM-5 criteria, including persistent depressive disorder with intermittent or persistent major depressive episode according to DSM-5, Premenstrual Dysphoric Disorder, Substance Induced Depressive Disorder, Depressive Disorder due to another Medical Condition, Other Specified or Unspecified Depressive Disorder, Bipolar Disorder I or II, depressed episode, Schizoaffective Disorder (Depressive or Bipolar type))
* Depression onset within 12 months after a stroke
* Suicidal risk defined as a score > 3 on the item 3 of the HAM-D scale or in the investigator's opinion
* Lactose intolerance
* Patients with hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Resistant depression for the current episode (patients who have not responded to 1 previous antidepressant treatment before the SSRI taken at an appropriate dose)
* Current panic disorder
* Obsessive compulsive disorder
* Current post traumatic stress disorder, current acute stress disorder
* Current or past psychotic disorder
* Any severe personality features

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2016-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HAM-D) total score expressed as change from baseline value | 8 weeks of treatment

SECONDARY OUTCOMES:
HAM-D total score | at week 0, week 2, week 4, week 6 and week 8
  Depressive symptoms
Response to treatment defined by HAM-D total score decrease from baseline ≥ 50% | at week 0, week 2, week 4, week 6 and week 8
  Depressive symptoms
Clinical Global Impression scale (CGI), item 1 (Severity of depression) and item 2 (global Improvement) scores, response to treatment (CGI item 2 = 1 or 2) | CGI item 1 at week 0, week 2, week 4, week 6 and week 8 and item 2 at week 2, week 4, week 6 and week 8
  Depressive symptoms
Hospital Anxiety and Depression Scale (HAD), Anxiety and Depression sub-scores | at week 0, week 2, week 4, week 6 and week 8
  Depressive symptoms
Sheehan Disability Scale (SDS) scores (Work, social and family life) | at week 0, week 2, week 4, week 6 and week 8
  Social functioning
Adverse Events | through study completion (an average of 12 weeks)
  Safety criterion
Body Weight | at week 4 and week 8
  Safety criterion
BMI | at week 4 and week 8
  Safety criterion
Laboratory tests (haematology and biochemistry) | at week 4 and week 8
  Safety criterion
12-lead ECG | at week 4 and week 8
  Safety criterion
Vital signs (standing and supine Systolic and Diastolic Blood Pressure, heart rate) | at week 0, week 2, week 4, week 6 and week 8
  Safety criterion
Columbia-Suicide Severity Rating Scale (C-SSRS) | at week 0, week 2, week 4, week 6 and week 8
  Safety criterion

CONTACTS AND LOCATIONS:
Locations (53):
- Bulgaria (6):
  - Mental Health Centre - Plovdiv, Plovdiv
  - Mental Health Centre - Sofia district, Sofia
  - Military Medical Academy, MHAT - Sofia, Sofia
  - Diagnostic Consultative center "Tchaika", Varna
  - Medical center "City clinic", Varna
  - Mental health centre - Vratsa, Vratsa
- Czechia (9):
  - Saint Anne s.r.o., Brno
  - Soukroma psychiatricka ambulance, Brno
  - Neuropsychiatrie HK, s.r.o., Hradec Králové
  - Bialbi s.r.o., Litoměřice
  - CLINTRIAL s.r.o., Prague
  - AD71 s.r.o., Prague
  - Pragtis s.r.o., Prague
  - Medical services Prague s.r.o., Prague
  - Psychiatricka ambulance Strakonice, Strakonice
- Finland (4):
  - Laakarikeskus Mehilainen Psychiatric, Helsinki
  - Private Practice, Kuopio
  - Oulu Mentalcare Oy, Research Unit, Oulu
  - Mentoria Oy, Tampere
- Hungary (10):
  - Bajai Szent Rokus Korhaz, Neurologia/Pszichiátria, Baja
  - Dr. Kenessey Albert Korhaz-Rendelointezet 1-es Pszihiatriai Osztaly, Balassagyarmat
  - Forras Outpatient Clinic, Budapest
  - Semmelweis Orvostudomanyi Egyetem, Pszichiatriai es Pszichoterapias Klinika, Budapest
  - Nyiro Gyula Korhaz, Pszihiatriai Osztaly, Budapest
  - Processus Kft., Városkapu Rendelo, Budapest
  - Petz Aladar Megyei Oktato Korhaz, Pszihiatriai, Mentalhygienes es Addiktologiai Osztaly, Győr
  - Bekes Megyei Pandy Kalman Korhaz, Pszihiatriai Osztaly, Gyula
  - Pecsi Tudomanyegyetem, Klinikai Kozpont, Pszich. es Pszichoter. Klinika, Pécs
  - Szent-Gyorgyi Albert Klinikai Kozpont, Pszichiatriai Klinika, Szeged
- Russia (7):
  - Psychiatric Hospital N 13, Moscow
  - Scientific Center of Mental Health, Dpt of Psychiatry N 1, Moscow
  - State Budgetary lnstitution of Healthcare Leningrad RPND, In-patient psychiatry department, Roshchino
  - Scientific Center for Treatment and Rehabilitation Phoenix, Research department, Rostov-on-Don
  - Psychoneuropathology Dispensary N 10, Psychiatry dpt, Saint Petersburg
  - City Psychiatric Hospital N 4, Psychiatric department, Saint Petersburg
  - V.M.Bekhterev Research Institute of Psychoneurology, Department of the neuroses and psychotherapy, Saint Petersburg
- Slovakia (7):
  - Psychiatricka ambulancia Mentum, s.r.o., Bratislava
  - VAVRUSOVA CONSULTING s.r.o., Nestatna psychiatricka ambulancia, Bratislava
  - INVESTA, spol. s r.o., Psychiatricka ambulancia, Košice
  - Private practice, Kysucké Nové Mesto
  - PsychoLine psychiatricka ambulancia s.r.o., Rimavská Sobota
  - NsP Svatej Barbory, Psychiatricke oddelenie, Rožňava
  - Centrum zdravia R.B.K. s.r.o., Svidník
- Ukraine (10):
  - Institute of Neurology, Psychiatry and Narcology, Department of Borderline and Neurotic Disorders, Kharkiv
  - Kherson Regional Psychiatric Hospital, Psychiatry department, Kherson
  - Kyiv Municipal Psychiatric Hospital #2, Department of psychiatry, Kyiv
  - Railway Clinic Hospital #1, Psychoneurological dpt, Kyiv
  - Kyiv Regional Medical Incorporation "Psychiatry", Center of Novel Treatment Rehabilitation Psychotic disorders, Kyiv
  - Ukrainian Research Institut of Social, Forensic Psyshiatry, Department of Therapy, Kyiv
  - Lviv District Psychiatric hospital, Lviv
  - Regional Clinic of Psychiatry, Lviv
  - ODESA REGIONAL MEDICAL CENTRE OF MENTAL HEALTHE DAY CARE department, Odesa
  - Odesa Regional Medical Centre of Mental Health Child-adolescens, Odesa

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/